CLINICAL TRIAL: NCT06050772
Title: Effect of Immersive Virtual Reality Reminiscence Versus Traditional Reminiscence Therapy on Cognitive Function and Psychological Wellbeing Among Institutionalized Older Adults: A Randomized Controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Mahmoud Khedr, Lecturer, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 71-d
Record Dates: First submitted 2023-09-17; First posted 2023-09-22 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Institutionalized Older Adults

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- STUDY GROUP (Experimental): Groups who will receive virtual reality reminiscence versus traditional reminiscence therapy to determine its effect on cognitive function and psychological wellbeing.
  Interventions: Behavioral: Immersive Virtual Reality Reminiscence; Behavioral: Traditional Reminiscence Therapy
- Control group (No Intervention): Groups who will not receive any intervention

INTERVENTIONS:
Behavioral: Immersive Virtual Reality Reminiscence — a computer-generated environment using head-mounted displays (HMDs) that provide a fully immersive, completely engaging, and realistic experience so that users feel like they are a part of the virtual world
  Arms: STUDY GROUP
Behavioral: Traditional Reminiscence Therapy — RT is a technique that encourages older adults' positive emotions and coping mechanisms by using the recall of earlier memories and the sharing of life experiences.
  Arms: STUDY GROUP

SUMMARY:
Cognitive function and psychological wellbeing are basic determinants of successful ageing that enable older adults to maintain their health, independence, and autonomy. Reminiscence therapy (RT) is one of the most prevalent evidence-based psychosocial interventions that can enhance older adults' cognitive function and maintain their psychological health. Virtual reality (VR) reminiscence is an innovative strategy that has the advantage of integrating technology in to the care of institutionalized older adults. However, limited researches have been conducted to compare the role of VR reminiscence versus traditional RT on improving older adult's cognitive and psychological wellbeing.

DETAILED DESCRIPTION:
The aim of this study is to determine the effect of virtual reality reminiscence versus traditional reminiscence therapy on cognitive function and psychological wellbeing among institutionalized older adults.

ELIGIBILITY:
Inclusion Criteria:

* their age is 60 years and above, capable of communicating clearly, free form hearing or vision impairments that might hinder RT, and being able to tolerate using the Head Mounted Display(HMD) headset.

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-03-20 (Actual); Primary Completion 2023-09-25 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
cognitive function | 3 months
  The Mini-Mental State Examination (MMS) is recommended as an effective predictor of cognitive function of the elderly people . It involves six cognitive related subscales with eleven questions investigating memory, concentration, orientation to time and place, registration, calculation, repetition, naming objects, language and recall.
Psychological Wellbeing | 3 months
  The PWB measures six dimensions of psychological wellbeing among older adults including autonomy, environmental mastery, personal development, supportive relationships, purpose in life, and acceptance of oneself
Virtual Reality | 3 months
  The CSQ-VR is a widely used scale to assess side effects of VR due to several advantages; it is easy applicable tool, it has clear questions and answers, its coring is simple and easy to understand, and its items cover all VR related symptoms.
Immersive Virtual Reality | 3 months
  This questionnaire was adapted from the User eXperience in Immersive Virtual Environment Questionnaire (UX in IVEQ). It was used to assess the participant's experience in immersive VR. It is made up of 16 items which are distributed across 5 domains including presence (4 items), engagement (3 items), immersion (3 item), flow (3 items), and emotion (3 items).

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Nursing, Damnhour university, Damanhūr, Egypt

IPD SHARING:
Plan to Share IPD: No